CLINICAL TRIAL: NCT06919250
Title: Physical Activity and Its Impact on Health in Patients With Systemic Lupus Erythematosus. A Multicenter Cohort Study.
Brief Title: Physical Activity in Patients With Systemic Lupus Erythematosus
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Ruben Cuesta Barriuso, Principal Investigator, University of Oviedo
Other Study IDs: ActLup
Record Dates: First submitted 2025-03-25; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Systemic Lupus Erythematosus; Physical activity; Prevention; Physiotherapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with systemic lupus erythematosus: Patients with systemic lupus erythematosus who will participate through an interview format with closed questions where no data will be collected that would allow identification of the subjects.
  Interventions: Other: Patients with systemic lupus erythematosus

INTERVENTIONS:
Other: Patients with systemic lupus erythematosus — Population: Patients with systemic lupus erythematosus. Intervention: Identification of the degree of physical activity of patients with systemic lupus erythematosus.

SUMMARY:
Background. Systemic lupus erythematosus is a chronic autoimmune disease. Among its main clinical manifestations are musculoskeletal symptoms such as myopathies, arthritis, arthralgias or osteonecrosis. Physical activity can improve the perception of quality of life and well-being of these patients.

Objective. To assess the degree of physical activity in patients with systemic lupus erythematosus, and to identify the main clinical, sociodemographic and anthropometric variables that influence it.

Method. Ambispective cohort study. Sixty-three patients with systemic lupus erythematosus will be recruited. The primary variable will be the degree of physical activity (International Physical Activity Questionnaire). Secondary and modifying variables will be: fatigue (Fatigue Assessment Scale), health-related quality of life (Short Form-36 Health Survey), sleep disorders (Pittsburgh Sleep Quality Index), depressive (Beck Depression Inventory -II) and anxiety symptoms (Hamilton Anxiety Rating Scale), age, and disease activity, duration and damage. Possible confounding variables will be sex, toxic habits (smoking), diagnosis of other pathologies and exposure to therapy. In the analysis, the degree of physical activity of patients with lupus erythematosus will be calculated and a multiple regression analysis will be performed to evaluate the predictive model that best fits the degree of activity of these patients.

Expectedresults. To identify the degree of physical activity of patients with systemic lupus erythematosus and to identify the predictive model of physical activity in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of systemic lupus erythematosus
* Of legal age
* Residents in Spain
* Who sign the informed consent document.

Exclusion Criteria:

* Patients dependent in the development of activities of daily living.
* Unable to ambulate without the help of third parties.
* Who have undergone surgery in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic lupus erythematosus
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of the degree of physical activity | Screening visit
  The degree of physical activity will be assessed with the International Physical Activity Questionnaire (IPAQ). This tool assesses the time spent walking and sitting. The results are classified into three categories: low, moderate and high activity. The unit of measurement is the units of measurement of the metabolic rate (METS), where the higher the number of METS, the greater the physical activity.

SECONDARY OUTCOMES:
Measurement of health-related quality of life | Screening visit
  Health-related quality of life will be measured with the Short Form-36 Health Survey questionnaire. It is composed of 36 items that inquire about 8 dimensions (physical function, physical role, bodily pain, general health, vitality, social function, emotional role, and mental health, including a health transition item). The score range is from 0 to 100 (best perception of quality of life).
Measurement of fatigue | Screening visit
  The degree of fatigue will be measured with the Fatigue Assessment Scale questionnaire. This instrument assesses perceived mental and physical fatigue, consisting of 10 items. The score varies between 10 and 50 points, where the higher the score the higher the level of fatigue.
Measurement of sleep disorders | Screening visit
  Sleep disorders will be measured with the Pittsburgh Sleep Quality Index. This questionnaire examines in 7 dimensions subjective sleep quality, sleep latency and duration, and sleep efficiency and disturbances, use of sleep medications, and daytime dysfunction. It is composed of 19 items. The score range varies from 0 to 21, considering poor sleep quality a score higher than 5 and good sleep quality if it is lower than 5 points
Measurement of depressive symptoms | Screening visit
  The depressive symptoms of the patients included in the study will be assessed with the Beck Depression Inventory. This tool consists of 21 items, grouped into 4 dimensions: emotional, cognitive, motivational and physiological. The scores vary between 0 and 63 points, and a state of absence or minimal depression (0-13 points), mild depression (14-19 points), moderate depression (20-28 points) or severe depression (29-63 points) can be obtained. A cut-off point of 15 points or more is proposed to diagnose depression.
Measurement of anxiety symptoms | Screening visit
  The Hamilton Anxiety Rating Scalewill be used to measure patients' anxiety symptoms. This scale quantifies the severity of anxiety by means of 14 items associated with somatic and psychological symptoms. Based on responses, patients are grouped into three categories: mild or absent anxiety (<17 points), mild-moderate (18 to 24 points) or moderate to severe (25-30 or more). The total score ranges from 0 to 56, where the higher the score, the greater the anxiety.
Measurement of age | Screening visit
  The measurement of age, a quantitative variable, will be made taking as a unit the number of years completed.
Measurement of disease activity | Screening visit
  The measurement of disease activity, a quantitative variable, will be made with the specific scale for patients with Systemic Lupus Erythematosus Disease Activity Index (SLEDAI), with a score from 0 to 105 points
Measurement of disease damage | Screening visit
  The measurement of disease damage, a quantitative variable, will be made with the specific scale for patients with lupus erythematosus sitematosus SLICC Damage Index (SDI), with a score of 0 to 46.
Measurement of disease duration | Screening visit
  Measurement of disease duration, a quantitative variable, will be calculated in months completed.

OTHER OUTCOMES:
Measurement of gender | Screening visit
  Gender, a dichotomous variable (Male/Female), will be a possible confounding variable.
Measurement of toxic habits | Screening visit
  Smoking as a toxic habit, dichotomous variable (Yes/No), will be a possible confounding variable.
Assessment of the diagnosis of other pathologies with a questionnaire | Screening visit
  The assessment of the diagnosis of other pathologies will be a possible confounding variable. In the evaluation questionnaire, patients will be able to indicate whether they have been diagnosed with another pathology, with this variable having multiple answers in those cases of patients with different pathologies.
Evaluation of the usual pharmacological treatment received by patients, by means of a specific question in a questionnaire | Screening visit
  The usual pharmacological treatment, a nominal qualitative polytomous variable (glucocorticoids / antimalarials / immunosuppressants), will be a possible confounding variable. This variable will be measured with the evaluation questionnaire, where patients will be able to respond with multiple answers.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Study Director — Universidad de Oviedo
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided